CLINICAL TRIAL: NCT03609411
Title: Splenectomy During Whole Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CRC_GHN_2018_002
Record Dates: First submitted 2018-07-17; First posted 2018-08-01 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: End Stage Liver Disease
MeSH Terms: conditions — End Stage Liver Disease | interventions — Splenectomy; Liver Transplantation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Splenectomy: Patients undergoing liver transplantation with simultaneous splenectomy
  Interventions: Procedure: Splenectomy
- Liver transplantation: Patients undergoing liver transplantation only

INTERVENTIONS:
Procedure: Splenectomy — Splenectomy was performed after hepatectomy, in an extra-hilar manner with manual ligation of splenic vessels.
  Other Names: Liver transplantation
  Groups: Splenectomy

SUMMARY:
Indications for splenectomy during whole liver transplantation remain controversial and splenectomy is often avoided because of common complications. The objective is to evaluate specific complications of these combined procedures.

DETAILED DESCRIPTION:
Data on patients who underwent splenectomy during liver transplantation were retrospectively analyzed . Participants underwent splenectomy as part of routine medical care. Patients undergoing simultaneous liver transplantation and splenectomy were matched to a non-splenectomy group.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing liver transplantation between 1994 and 2013

Exclusion Criteria:

* Data from living donor patients, split liver transplantation, patients with pre- or post-operative splenectomy in medical history, and patients under 16 years were excluded from analysis

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Among the 906 liver transplantations performed between 1994 and 2013 at the Liver Transplant Department of the Croix-Rousse University Hospital, Lyon-France, all 47 liver transplantations with simultaneous splenectomy were included and compared to 94 transplant recipients without splenectomy after a 1:2 matching for gender, age at transplantation, year of liver transplantation, MELD score, platelet level and presence of hepatocellular carcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
3-month post-operative mortality | At 3 months post surgery

SECONDARY OUTCOMES:
Post-operative morbidity | 3 months post surgery
  Incidence of portal-vein thrombosis within 3 months post liver transplantation
One-year mortality | One year after surgery
Mortality at 5 years | Five years after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital de la Croix-Rousse, Lyon, France

IPD SHARING:
Plan to Share IPD: No